CLINICAL TRIAL: NCT00863278
Title: Treatment of Melasma With Stabilized Kligman Preparation Associated or Not With Pulsed Dye Laser; a Comparative Prospective Study
Brief Title: Treatment of Melasma With Stabilized Kligman Preparation Associated or Not With Pulsed Dye Laser
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-PP-13
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2009-06

CONDITIONS: Melanosis
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): All patients will be treated by stabilized Kligman's trio with daily application during 4 months.
  After one month, the left side of the face will be treated with pulsed dye laser at the rate of 3 sessions (one every weeks).
  Applications of cream will be stopped on both side of the face for the 3 days following each laser session. Final visit will be scheduled 1 month after the end of applications of stabilized Kligman's trio.
  All the patients will used a sunscreen indication 50 + for the duration of the entire study.
  The patient is her own witness. They compare the hemiface treated without laser and the hemiface treated with the laser.
  Interventions: Procedure: pulsed dye laser treatment; Drug: Kligman's Trio
- Arm B (Active Comparator): All patients will be treated by stabilized Kligman's trio at the rate of application in the evening during 4 months.
  After one month, the side of the right face will be treated by pulsed dye laser at the rase of 3 sessions spaced out by 3 weeks each.
  Applications will be stopped in the 3 days which will follow every session by laser with blown colouring agent. The patients will be seen again 1 month after the stopping of applications of stabilized Kligman's trio
  All patients will be used a sunscreen indication 50 + for the duration of study.
  The patient is her own witness. They compare the cheek treated without laser and the cheek treated with the laser.
  Interventions: Procedure: pulsed dye laser treatment; Drug: Kligman's Trio

INTERVENTIONS:
Procedure: pulsed dye laser treatment — On one side of the face according to Arm placement.
Drug: Kligman's Trio — The combination of hydroquinone, retinoic acid and steroids combined in topical daily application.

SUMMARY:
Melasma is an acquired disorder of pigmentation that leads to irregular pigmented patches on the face. Treatment is difficult and to date the best treatment option is the combination of hydroquinone, retinoic acid and steroids combined in topical daily application (called Kligman's trio). Q-switched pigmentary lasers are usually ineffective and can induce post inflammatory hyperpigmentation (PIH). Intense pulsed light can sometimes improve melasma but also induce PIH which limit their use. Recently, pulsed dye laser were demonstrated to be effective in treating some pigmentary defects. Associating blanching cream with hydroquinone to prevent PIH after laser or intense pulsed light has been already reported with success.

The objective of the study is to compare in a prospective intra individual comparative trial the association of pulsed dye laser plus stabilized Kligman's trio to Kligman's trio alone. The secondary objective was to study the frequency and the intensity of the potential side effects including PIH.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women or breastfeeding.
* Skin type 5 or 6.

Exclusion Criteria:

* Known allergy to the compounds of the Kligman preparation.
* Refusal to put very high protection sunscreen during the study.
* Concomitant use of topical products that might have an effect on melasma (topical steroids, retinoids, etc…)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
MASI score, standardized photos in direct, crossed polarized and UV light, relating to the security: 0 yes 1 N0 | visit of screening (V0), 15 days after V0 during the follow visit 1(V1), 3 weeks after V1 during the following visit 2(V2), 3 weeks after V2 during the following visit 3(V3), 10 weeks after V3 during the following visit 4

SECONDARY OUTCOMES:
Clinical evaluation of potential side-effects (including post inflammatory pigmentation) | visit of screening (V0), 15 days after V0 during the follow visit 1(V1), 3 weeks after V1 during the following visit 2(V2), 3 weeks after V2 during the following visit 3(V3), 10 weeks after V3 during the following visit 4

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Ph Thierry, MD, Principal Investigator — CHU de Nice - Service de Dermatologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France